CLINICAL TRIAL: NCT06688942
Title: Digital Health Intervention to Promote Quality of Life in Adults With Chronic Graft Versus Host Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Lara Traeger, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20240864
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-12

CONDITIONS: Chronic Graft-Versus-Host Disease; Quality of Life
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Horizons Digital Health Application Group (Experimental): Participants will receive the Horizons mobile application for up to 6 weeks.
  Interventions: Behavioral: Horizons App Intervention

INTERVENTIONS:
Behavioral: Horizons App Intervention — Participants will receive access to the Horizons app intervention. The intervention pairs patient-centered information about chronic graft-versus-host disease with self-management strategies. Within each module, patients will engage in didactics and exercises that are relevant to the participant's chronic graft-versus-host disease concerns. The app contains 6 digital modules delivered via tablet over approximately 6 weeks. Each module should take up to approximately 20 minutes and are self-guided.

SUMMARY:
The goal of this interventional study is to learn if the Horizons mobile application is feasible for survivors of allogeneic hematopoietic stem cell transplant who have chronic graft-versus-host disease. Participants will be asked to complete surveys and use the Horizons mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Underwent allogeneic hematopoietic stem cell transplant
* Have moderate to severe chronic graft-versus-host disease
* Currently receiving care at the Sylvester Comprehensive Cancer Center Bone Marrow Transplant Program
* Able to use an Ipad to participate in the Horizons app intervention
* Able to participate in study procedures in English

Exclusion Criteria:

* comorbid conditions or cognitive impairment that the treating clinician believes prohibits informed consent or participation in the intervention
* Vulnerable patients, defined here as prisoners and pregnant women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Percentage of participant enrollment | Up to 8-week follow-up
  Participant enrollment will be demonstrated if ≥60% eligible participants enroll.
Percentage of participant retention | Up to 8-week follow-up
  Participant retention will be demonstrated if ≥80% participants are retained in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Traeger, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No